CLINICAL TRIAL: NCT05416684
Title: A Real World Prospective Observational Study on Evaluation the Comprehensive Effects of Polyetheretherketone Cranioplasty and Titanium Cranioplasty After Decompressive Craniectomy
Brief Title: Prospective Observational Study on Comprehensive Effects of PEEK Cranioplasty and Titanium Cranioplasty After DC（RECEPT-DC）
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Junfeng Feng, Director of Brain Injury Center, RenJi Hospital
Other Study IDs: IIT-2021-0111
Record Dates: First submitted 2022-05-28; First posted 2022-06-13 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Skull Defect
Keywords: Skull Defect; Epilepsy; Infections
MeSH Terms: conditions — Epilepsy; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PEEK Group
- Titanium Mesh Group

SUMMARY:
The objective of this trial is to scientifically evaluate the efficacy of PEEK cranioplasty and titanium cranioplasty. The primary objective is to compare the rate of implant failure (defined as infection, implant exposure and other causes requiring removal of the implanted material) at any time within 12 months after cranioplasty. The secondary objective is to compare the complication rates and neurological function recover following cranioplasty. Complication events after cranioplasty are investigated within 6 months after surgery and neurological function is evaluated at 3, 6 and 12 months after cranioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Skull defect with a diameter greater than 3cm
* No intracranial hemorrhage, intracranial hypertension or hydrocephalus (or treated) occurred more than 1 month after the previous operation
* Cranioplasty is feasible according to doctor's evaluation
* Patients must agree to participate in this clinical trial and the informed consent is signed by patients themselves or next of kin on behalf of the patient.

Exclusion Criteria:

* Manifestations of intracranial hypertension or untreated hydrocephalus
* Poor healing of skin wound
* Intracerebral infection or intracerebral hematoma is not cured
* Patients with operational contradictions, for example, poor general condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with skull defect
Sampling Method: Non-Probability Sample
Enrollment: 358 (Estimated)
Dates: Start 2024-11-07 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Implant Failure | Within 12 months
  implant failure (defined as infection, implant exposure and other causes requiring removal of the implanted material) at any time within 12 months after cranioplasty.

SECONDARY OUTCOMES:
Length of stay in hospital | Within 2 months post-operation
  The duration of hospitalization after operation.
Detailed Economic Evaluation | Within 6 months post-operation
  Total medical expense related to treatment of cranioplasty, including the costs of operations and hospitalization within 6 months post-injury.
Complications Rates | 3, 6, and 12 months
  including seizure, hematoma, hydrocephalus, etc.
Glasgow coma scale (GCS) | 3, 6, and 12 months
  The Glasgow coma scale (GCS) is used to assess and calculate the patient's level of consciousness.
Glasgow outcome scale (GOS) | 3, 6, and 12 months
Mini-Mental State Examination score (MMSE) | 3, 6, and 12 months
Appearance Satisfaction | 6 months
  Questionnaire was used to investigate patients' satisfaction with the appearance of cranioplasty.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China